CLINICAL TRIAL: NCT05643690
Title: Urine Sample Collection for Validation of the AnchorDx UriFind™ Bladder Cancer Assay in Subjects Suspected of Having Bladder Cancer
Brief Title: Urine Sample Collection for Validation of the AnchorDx UriFind™ Bladder Cancer Assay
Status: Suspended | Type: Observational
Why Stopped: Protocol amendment.
Sponsor: AnchorDx Medical Co. Ltd. US (Industry)
Collaborators: AnchorDx Medical Co., Ltd. (Industry); Specialty Networks (Unknown)
Responsible Party: Sponsor
Other Study IDs: UriFind US-001
Record Dates: First submitted 2022-11-14; First posted 2022-12-09 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Clinical Validation Group: Patients with suspected bladder cancer (including hematuria, inflammatory bladder, suspicious ultrasound results)
  Interventions: Diagnostic Test: UriFind Bladder Cancer Assay

INTERVENTIONS:
Diagnostic Test: UriFind Bladder Cancer Assay — The AnchorDx UriFind™ Bladder Cancer Assay is designed to detect 2 DNA methylation biomarkers in urine specimens from patients 22 years or older suspected of having bladder cancer. Results from the Assay are intended for use, in conjunction with current standard diagnostic procedures, as an aid for initial diagnosis of bladder carcinoma in patients.

SUMMARY:
The AnchorDx UriFind™ Bladder Cancer Assay is designed to detect 2 DNA methylation biomarkers in urine specimens from patients 22 years or older suspected of having bladder cancer. Results from the assay are intended for use, in conjunction with current standard diagnostic procedures, as an aid for initial diagnosis of bladder carcinoma in patients.

ELIGIBILITY:
Inclusion Criteria:

Clinical Validation Group:

1. 55 years or older, gender is not limited
2. Suspected of bladder cancer and are scheduled for bladder biopsy or trans-uretheral resection of bladder tumor (TUBRT)
3. Can receive standard of care, including urine cytology, cystoscopy, or surgery for bladder cancer diagnosis
4. Can provide at least of 75 ml of urine (prior to cystoscopy or surgery)

Exclusion Criteria:

1. History of urinary cancer
2. Neoadjuvant therapy

Ages: 55 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The clinical validation group is to assess the safety and effectiveness of the AnchorDx UriFind™ Bladder Cancer Assay in an intended use population to establish the expected performance in the product labeling. The study also aims to provide performance evidence of the AnchorDx UriFind™ Bladder Cancer Assay in adequate number of early-stage and low-grade cases.
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2022-11-18 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and Specificity of UriFind assay in detecting early stage Bladder Cancer | Baseline
  To evaluate the performance of the UriFind assay relative to the patient at diagnosis (cystoscopy or surgery followed by histology).

CONTACTS AND LOCATIONS:
Overall Officials: Jianbing Fan, Ph.D, Study Director — AnchorDx Medical Co., Ltd.
Locations (2):
- United States (2):
  - Arkansas Urology, Little Rock, Arkansas
  - Idaho Urologic Institute, Meridian, Idaho

IPD SHARING:
Plan to Share IPD: No